CLINICAL TRIAL: NCT05394038
Title: Application of Rapid Risk Stratification for Patients Presenting With Chest Pain in the Emergency Department During the Covid-19 Outbreak in Shanghai, China.
Brief Title: Rapid Diagnosis of Patients With Chest Pain During the Covid-19 Outbreak (My-ABCDE)
Acronym: My-ABCDE
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, Director, Director of Cardiovascular Medicine, Shanghai 10th People's Hospital
Other Study IDs: My-ABCDE
Record Dates: First submitted 2022-05-25; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Chest Pain
MeSH Terms: conditions — Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CPC Cohort: A patient with chest tightness and pain during the Covid-19 outbreak.
  Interventions: Other: None，observational study.

INTERVENTIONS:
Other: None，observational study. — observational study

SUMMARY:
During the outbreak of COVID-19, among patients with chest tightness and chest pain as the main symptoms in major medical institutions in Shanghai, China, the past medical history and rapid testing were used to quickly identify the risk stratification of the patients.

DETAILED DESCRIPTION:
During the outbreak of COVID-19, among patients with chest tightness and chest pain as the main symptoms in major medical institutions in Shanghai, China, the past medical history and rapid testing were used to quickly identify the risk stratification of the patients. Past medical history collection includes diabetes, hypertension, coronary atherosclerotic heart disease, percutaneous coronary stent implantation, etc. Rapid detection includes rapid myocardial markers, coagulation function, electrocardiogram, chest CT, etc. Risk stratification in the shortest possible time to reduce the time patients spend congregating in hospitals and reduce unnecessary contact to reduce the risk of Covid-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients who came to the hospital with chest tightness and chest pain during Covid-19.

Exclusion Criteria:

* None.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who came to the hospital with chest tightness and chest pain during Covid-19.
Sampling Method: Non-Probability Sample
Enrollment: 2218 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Diagnosis time | 1 week
  The time from the first medical contact to the time of diagnosis.

SECONDARY OUTCOMES:
Diagnostic accuracy | 1week
  Preliminary and confirmed diagnoses were the same proportion of the total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Yawei Xu, PhD, Study Chair — Tongji University
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No